CLINICAL TRIAL: NCT03259763
Title: EUS-guided Gastroenterostomy Versus Enteral Stenting for Palliation of Malignant Gastric Outlet Obstruction: A Randomized Clinical Trial
Brief Title: EUS-GE vs ES for Palliation of Gastric Outlet Obstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00128878
Record Dates: First submitted 2017-08-15; First posted 2017-08-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Gastric Outlet Obstruction
Keywords: Gastroenterostomy; Gastric Outlet Obstruction; Cancer; Endosonography
MeSH Terms: conditions — Gastric Outlet Obstruction; Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated with a 1:1 ratio to one of the study arms (EUS-GE or ES)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUS-guided gastroenterostomy (EUS-GE) (Active Comparator): In this technique, the gastric wall and its adjacent small intestine are punctured by a needle to make a connection between the stomach and small intestine. Then a lumen-apposing metal stent is deployed at the puncture site to keep the stomach-small intestine connection open.
  Interventions: Device: Lumen-apposing metal stent
- Enteral Stenting (ES) (Active Comparator): In this technique, under endoscopic visualization, a guidewire will be advanced through the obstructed part of the stomach. Then an enteral self-expandable metal stent will be deployed under direct endoscopic visualization and fluoroscopic guidance.
  Interventions: Device: Self-expandable metal stent

INTERVENTIONS:
Device: Lumen-apposing metal stent — In this technique, the gastric wall and its adjacent small intestine are punctured by a needle to make a connection between the stomach and small intestine. Then a lumen-apposing metal stent is deployed at the puncture site to keep the stomach-small intestine connection open.
  Arms: EUS-guided gastroenterostomy (EUS-GE)
Device: Self-expandable metal stent — In this technique, under endoscopic visualization, a guidewire will be advanced through the obstructed part of the stomach. Then an enteral self-expandable metal stent will be deployed under direct endoscopic visualization and fluoroscopic guidance.
  Arms: Enteral Stenting (ES)

SUMMARY:
Gastric outlet obstruction (GOO) is a common complication of luminal malignancies which is associated with substantial morbidity. Palliation of GOO has traditionally been through the surgical bypass of the obstructed lumen by creating an opening between the stomach and small intestine. However, In recent years, a less invasive approach, i.e. endoscopic stenting, has gained wide acceptance to treat unresectable malignant gastric outlet obstruction. In this study, the investigators are going to compare the safety and efficacy of the two different endoscopic techniques including Endoscopic ultrasonography-guided gastroenterostomy (EUS-GE) and enteral stenting (ES).

DETAILED DESCRIPTION:
In recent years, Enteral Stenting (ES) has commonly been used as the first line management of unresectable malignant gastric outlet obstruction. On the other hand, Endoscopic ultrasonography-guided gastroenterostomy (EUS-GE) is the most recently described technique for palliation of malignant GOO, which has the theoretical potential to minimize the risk for stent occlusion while maintaining the less invasive endoscopic approach. This novel endoscopic treatment entails creating a gastroenterostomy under EUS-guidance thereby bypassing the occluded lumen. This endoscopic technique has been performed to treat patients with GOO since 2014, and recent retrospective studies have shown that EUS-GE was comparable to ES in terms of efficacy and safety; however, EUS-GE was associated with a significantly decreased risk of recurrent GOO and reinterventions.

Based on the investigator's clinical experience for the last three years and the above-mentioned study results, the goal of this study is to prospectively compare EUS-GE with ES in the management of unresectable malignant gastric outlet obstruction. The investigators hypothesize that EUS-GE is associated with comparable technical and clinical success and safety profile while requiring fewer re-interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with malignant, symptomatic gastric outlet obstruction due to an unresectable malignant lesion
* Gastric outlet obstruction scoring system (GOOSS) score of 0 (no oral intake) or 1 (liquids only)
* Age 18-80 years

Exclusion Criteria:

* Evidence of other strictures in the gastrointestinal (GI) tract
* Previous gastric, periampullary or duodenal surgery
* World Health Organization (WHO) performance score of 4 (patient is 100% of time in bed)
* Unable to fill out quality of life questionnaire
* Unable to sign the informed consent
* Life expectancy of less than 3 months based on the endoscopist's opinion
* Cancer extending into the body of the stomach, 4th portion of the duodenum or proximal jejunum around the ligament of Treitz
* Large volume ascites
* Inability to tolerate sedated upper endoscopy due to cardiopulmonary instability, severe pulmonary disease or other severe comorbidities
* Pregnant or breastfeeding women
* Uncorrectable coagulopathy defined by INR > 1.5 or platelet < 50000/µl
* Complete GOO evidenced by inability to either pass a wire across the stricture and/or inability to opacify small bowel distal to the malignant stricture
* Resectable or borderline resectable tumors
* One of the two techniques (EUS-GE and ES) cannot be performed (at the discretion of the endoscopist)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Rate of gastric outlet obstruction recurrence | 3 months
  Recurrence of nausea, vomiting, and inability to tolerate PO intake up to 3 months after the procedure confirmed either endoscopically and/or radiographically.

SECONDARY OUTCOMES:
Technical success rate | Day of procedure
  Adequate positioning and deployment of the stent(s) as determined endoscopically and radiographically.
Clinical success rate | 1 week
  The improvement of at least 1 point in the gastric outlet obstruction score within 7 days after stent insertion.
Length of procedure | Day of procedure
Adverse events rate | 1 week
Post-procedure length of hospital stay | 1 week
Reintervention rate for recurrent gastric outlet obstruction | 3 months
Quality of Life SF-36 questionnaire scoring | 3 months
  The SF-36 general health questionnaire consists of 36 questions evaluating the patient's perception of their quality of life (QoL) in the following eight subscales: physical functioning (PF), role limitations due to physical problems (RP), role limitations due to emotional problems (RE), energy/fatigue (EF), emotional well-being (EW), social functioning (SF), bodily pain (BP) and general health (GH). Subscale scores range from 0 to 100, with 100 being the best and 0 being the worst quality of life.
Overall survival rate | 1 year
Time to recurrent gastric outlet obstruction | 3 months
Gastric Outlet Obstruction Scoring system (GOOSS) | 1 year
  Diet toleration will be scored based on the Gastric Outlet Obstruction Scoring System (GOOSS). The scoring ranges from 0 to 3 in the following format:
  0 = no oral intake, 1 = liquids only, 2 = soft solids, 3 = low-residue or full diet
Stent Dysfunction Rate | 3 months
  the restenosis of the stent due to tumor ingrowth or overgrowth, stent migration, or fracture
Duration of stent patency | 3 months
  Calculated from the time of stent placement to the time of stent dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A. Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (3):
  - Yale University, New Haven, Connecticut
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Wake Forest Baptist University, Winston-Salem, North Carolina
- The Research Institute of McGill University Health Centre, Montreal, Quebec, Canada
- Ecuadorian Institute of Digestive Diseases (IECED), Guayaquil, Ecuador
- Hospital Prive des Peupliers, Paris, France
- Asian Institute of Gastroenterology, Hyderabad, India
- Emek Medical Center, Afula, Israel
- Hospital Universitario Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittal A, Windsor J, Woodfield J, Casey P, Lane M. Matched study of three methods for palliation of malignant pyloroduodenal obstruction. Br J Surg. 2004 Feb;91(2):205-9. doi: 10.1002/bjs.4396. PMID 14760669
- [Background] Johnsson E, Thune A, Liedman B. Palliation of malignant gastroduodenal obstruction with open surgical bypass or endoscopic stenting: clinical outcome and health economic evaluation. World J Surg. 2004 Aug;28(8):812-7. doi: 10.1007/s00268-004-7329-0. Epub 2004 Aug 3. PMID 15457364
- [Background] Maetani I, Akatsuka S, Ikeda M, Tada T, Ukita T, Nakamura Y, Nagao J, Sakai Y. Self-expandable metallic stent placement for palliation in gastric outlet obstructions caused by gastric cancer: a comparison with surgical gastrojejunostomy. J Gastroenterol. 2005 Oct;40(10):932-7. doi: 10.1007/s00535-005-1651-7. PMID 16261429
- [Background] Khashab M, Alawad AS, Shin EJ, Kim K, Bourdel N, Singh VK, Lennon AM, Hutfless S, Sharaiha RZ, Amateau S, Okolo PI, Makary MA, Wolfgang C, Canto MI, Kalloo AN. Enteral stenting versus gastrojejunostomy for palliation of malignant gastric outlet obstruction. Surg Endosc. 2013 Jun;27(6):2068-75. doi: 10.1007/s00464-012-2712-7. Epub 2013 Jan 9. PMID 23299137
- [Background] Khashab MA, Kumbhari V, Grimm IS, Ngamruengphong S, Aguila G, El Zein M, Kalloo AN, Baron TH. EUS-guided gastroenterostomy: the first U.S. clinical experience (with video). Gastrointest Endosc. 2015 Nov;82(5):932-8. doi: 10.1016/j.gie.2015.06.017. Epub 2015 Jul 26. PMID 26215646
- [Background] Itoi T, Baron TH, Khashab MA, Tsuchiya T, Irani S, Dhir V, Bun Teoh AY. Technical review of endoscopic ultrasonography-guided gastroenterostomy in 2017. Dig Endosc. 2017 May;29(4):495-502. doi: 10.1111/den.12794. Epub 2017 Jan 27. PMID 28032663
- [Background] Chen YI, Itoi T, Baron TH, Nieto J, Haito-Chavez Y, Grimm IS, Ismail A, Ngamruengphong S, Bukhari M, Hajiyeva G, Alawad AS, Kumbhari V, Khashab MA. EUS-guided gastroenterostomy is comparable to enteral stenting with fewer re-interventions in malignant gastric outlet obstruction. Surg Endosc. 2017 Jul;31(7):2946-2952. doi: 10.1007/s00464-016-5311-1. Epub 2016 Nov 10. PMID 27834024
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Adler DG, Baron TH. Endoscopic palliation of malignant gastric outlet obstruction using self-expanding metal stents: experience in 36 patients. Am J Gastroenterol. 2002 Jan;97(1):72-8. doi: 10.1111/j.1572-0241.2002.05423.x. PMID 11808972